CLINICAL TRIAL: NCT02903537
Title: Tolerance-Induction With Dendritic Cells Treated With Vitamin-D3 and Loaded With Myelin Peptides, in Multiple Sclerosis Patients (TOLERVIT-MS)
Brief Title: Tolerogenic Dendritic Cells as a Therapeutic Strategy for the Treatment of Multiple Sclerosis Patients (TOLERVIT-MS)
Acronym: TOLERVIT-MS
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fundació Institut Germans Trias i Pujol (Other)
Collaborators: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TOLERVIT-MS; 2015-003541-26 (EudraCT Number)
Record Dates: First submitted 2016-07-21; First posted 2016-09-16 (Estimated); Last update posted 2023-07-07 (Actual); Status verified 2023-07

CONDITIONS: Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive
Keywords: Multiple Sclerosis; Dendritic Cells; Immune Tolerance; Myelin Proteins; Tolerogenic dendritic cells
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis, Chronic Progressive; Multiple Sclerosis | interventions — Interferon-beta

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 5 * 10 ^6 tolDC-VitD3 (Experimental): 5 million autologous VitD3 tolerogenic monocyte-derived dendritic cells loaded with a pool of myelin peptides (tolDC-VitD3)
  Interventions: Drug: Autologous VitD3 tolerogenic monocyte-derived dendritic cells loaded with a pool of myelin peptides (tolDC-VitD3)
- 10 * 10 ^6 tolDC-VitD3 (Experimental): 10 million autologous VitD3 tolerogenic monocyte-derived dendritic cells loaded with a pool of myelin peptides (tolDC-VitD3).
  Interventions: Drug: Autologous VitD3 tolerogenic monocyte-derived dendritic cells loaded with a pool of myelin peptides (tolDC-VitD3)
- 15 * 10 ^6 tolDC-VitD3 (Experimental): 15 million autologous VitD3 tolerogenic monocyte-derived dendritic cells loaded with a pool of myelin peptides (tolDC-VitD3).
  Interventions: Drug: Autologous VitD3 tolerogenic monocyte-derived dendritic cells loaded with a pool of myelin peptides (tolDC-VitD3)
- Interferon-beta (Experimental): Additional group (patients treated with beta-interferon) will receive the selected dose of those 3 previously cohorts studied
  Interventions: Drug: Autologous VitD3 tolerogenic monocyte-derived dendritic cells loaded with a pool of myelin peptides (tolDC-VitD3); Drug: Interferon-beta

INTERVENTIONS:
Drug: Autologous VitD3 tolerogenic monocyte-derived dendritic cells loaded with a pool of myelin peptides (tolDC-VitD3) — Intranodal administration
  Other Names: tolDC-VitD3
Drug: Interferon-beta — Subcutaneous administration interferon-beta
  Other Names: beta-interferon
  Arms: Interferon-beta

SUMMARY:
The purpose of this study is to determine the safety and tolerability of the intranodal administration of autologous monocyte-derived dendritic cells tolerised with Vitamin-D3 and pulsed with myelin peptides (tolDC-VitD3) in multiple sclerosis patients . To select the most appropriate regime for the development of future therapeutic trials.

To evaluate the preliminary proof of concept by clinical and/or radiological activity and immunological markers.

DETAILED DESCRIPTION:
Phase I dose ascending ("best of five") clinical trial.

First group will start by intranodal injection in cervical lymph nodes of 5*10^6 tolDC-VitD3.

Up titration depending on security outcomes to 10*10^6 tolDC-VitD3, same route in second cohort dose and next uptitration to 15*10^6 tolDC-VitD3.

Six cycles per patient with the following schema: for the first four cycles the administration will be each 2 weeks, for the remaining 2 cycles administration each 4 weeks.

A last cohort with the dose identified in the previous groups, administered in patients treated with beta interferon, same route, same dose schema.

ELIGIBILITY:
Inclusion Criteria:

1. EDSS of 0.0 - 6.5.
2. Multiple Sclerosis according to 2010 revised Mc Donald criteria, and less than 15 years of evolution of disease.
3. Patients with:

   * Active relapsing remitting multiple sclerosis (RRMS) (more than 1 relapse in last year and/or occurrence of ≥3 new T2 lesions or Gd positive) who not wish to be treated with current therapies.
   * Low activity RRMS (1 relapse in last year or occurrence of 1 or 2 T2 lesions or Gd positive) without treatment.
   * Progressive forms of MS with activity (at least 1 relapse in last year or occurrence 1 or 2 T2 lesions or Gd positive).
   * RRMS treated with interferon beta (Additional group)
4. T cell proliferation to the pool of myelin peptides against which is to induce immune tolerance: Myelin basic protein (MBP)13-32, MBP83-99, MBP111-129, MBP146-170, proteolipid protein (PLP) 139-154, Myelin oligodendrocyte glycoprotein (MOG)1-20, MOG35 -55).
5. Adequate peripheral venous access.
6. Signed informed consent.

Exclusion Criteria:

1. Use of corticosteroids during the prior 4 weeks.
2. Use of interferon beta -in patients who is retired by inefficiency or other causes- and glatiramer acetate in the 4 weeks prior.
3. Use of fingolimod, dimethylfumarate, natalizumab, immunoglobulins or plasmapheresis at 12 weeks; and teriflunomide in the 15 weeks prior.
4. Use of azathioprine, mitoxantrone, rituximab, methotrexate, cyclophosphamide, cyclosporine, alemtuzumab or other immunosuppressive drug, except corticosteroids, at any time.
5. Bone marrow or stem cell transplant at any time.
6. Relapse during the month prior of starting treatment. If it appears and the patient meets the eligibility criteria, must wait long enough until the end of the 30 days free of relapse. If corticosteroids are administered, the MRI performed during this period should not be considered, and a new MRI will be performed at 4 weeks after administration of corticosteroids.
7. Pregnancy or planning pregnancy within the next 12 months and breastfeeding.
8. Fertile patients who are not using an appropriate method of contraception. If the patient is menopausal or sterile it must be documented in the medical record.
9. Abusing drugs or alcohol.
10. Inability to undergo MRI evaluations.
11. Seropositivity for HIV, hepatitis B or C and/or syphilis.
12. History of oncological disease.
13. Clinically relevant concomitant disease: cardiac, pulmonary, neurological, renal or other major illness.
14. Splenectomy.
15. Dementia, psychiatric problems or other comorbidities that might interfere protocol compliance.
16. To be participating in another clinical study or to have participated in one in the last 3 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Estimated)
Dates: Start 2017-07-06 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Safety as assessed by the occurrence and severity of adverse events | 24 months
  Occurence and severity of adverse events will be recorded
Neurologic changes | 24 months
  New relapse. Disability progression on Expanded Disability Status Scale (EDSS)
Radiologic changes | 24 months
  Number of new or enlarging T2 lesions on brain MRI. Number of Gadolinium (Gd)-enhancing T1 lesions on brain MRI

SECONDARY OUTCOMES:
Annual relapse rate (ARR) | 24 months
Expanded Disability Status Scale (EDSS) | 24 months
9-Hole Peg Test (9HPT) | 24 months
25-Foot Walking Test (T25FW) | 24 months
Symbol Digit Modalities Test (SDMT) | 24 months
Radiologic preliminary efficacy | 24 months
  Number of new or enlarging T2 lesions on brain MRI. Number of Gadolinium (Gd)-enhancing T1 lesions on brain MRI
Lymphocyte proliferation to myelin peptides | 24 months
Blood Immunomonitoring studies | 24 months
Feasibility | 6 months
  Generation of Good Manufacturing Practices (GMP)-grade cell product released according to Quality Control. Feasibility of cellular product injection.

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Ramo, MD.PhD.Neurologist, Principal Investigator — Badalona Hospital Germans Trias i Pujol. Neurology service. Multiple Sclerosis department; Eva Martínez-Cáceres, MD.PhD.Immunology, Study Director — Badalona Hospital Germans Trias i Pujol. Immunology
Locations (2):
- Spain (2):
  - Hospital Universitari Germans Trias i Pujol, Badalona, Barcelona
  - Clínica Universidad de Navarra, Pamplona, Navarre

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lutterotti A, Yousef S, Sputtek A, Sturner KH, Stellmann JP, Breiden P, Reinhardt S, Schulze C, Bester M, Heesen C, Schippling S, Miller SD, Sospedra M, Martin R. Antigen-specific tolerance by autologous myelin peptide-coupled cells: a phase 1 trial in multiple sclerosis. Sci Transl Med. 2013 Jun 5;5(188):188ra75. doi: 10.1126/scitranslmed.3006168. PMID 23740901
- [Background] Giannoukakis N, Phillips B, Finegold D, Harnaha J, Trucco M. Phase I (safety) study of autologous tolerogenic dendritic cells in type 1 diabetic patients. Diabetes Care. 2011 Sep;34(9):2026-32. doi: 10.2337/dc11-0472. Epub 2011 Jun 16. PMID 21680720
- [Background] Benham H, Nel HJ, Law SC, Mehdi AM, Street S, Ramnoruth N, Pahau H, Lee BT, Ng J, Brunck ME, Hyde C, Trouw LA, Dudek NL, Purcell AW, O'Sullivan BJ, Connolly JE, Paul SK, Le Cao KA, Thomas R. Citrullinated peptide dendritic cell immunotherapy in HLA risk genotype-positive rheumatoid arthritis patients. Sci Transl Med. 2015 Jun 3;7(290):290ra87. doi: 10.1126/scitranslmed.aaa9301. PMID 26041704
- [Background] Naranjo-Gomez M, Raich-Regue D, Onate C, Grau-Lopez L, Ramo-Tello C, Pujol-Borrell R, Martinez-Caceres E, Borras FE. Comparative study of clinical grade human tolerogenic dendritic cells. J Transl Med. 2011 Jun 9;9:89. doi: 10.1186/1479-5876-9-89. PMID 21658226
- [Background] Raiotach-Regue D, Grau-Lopez L, Naranjo-Gomez M, Ramo-Tello C, Pujol-Borrell R, Martinez-Caceres E, Borras FE. Stable antigen-specific T-cell hyporesponsiveness induced by tolerogenic dendritic cells from multiple sclerosis patients. Eur J Immunol. 2012 Mar;42(3):771-82. doi: 10.1002/eji.201141835. PMID 22488365
- [Background] Mansilla MJ, Selles-Moreno C, Fabregas-Puig S, Amoedo J, Navarro-Barriuso J, Teniente-Serra A, Grau-Lopez L, Ramo-Tello C, Martinez-Caceres EM. Beneficial effect of tolerogenic dendritic cells pulsed with MOG autoantigen in experimental autoimmune encephalomyelitis. CNS Neurosci Ther. 2015 Mar;21(3):222-30. doi: 10.1111/cns.12342. Epub 2014 Nov 18. PMID 25403984
- [Background] Raich-Regue D, Naranjo-Gomez M, Grau-Lopez L, Ramo C, Pujol-Borrell R, Martinez-Caceres E, Borras FE. Differential effects of monophosphoryl lipid A and cytokine cocktail as maturation stimuli of immunogenic and tolerogenic dendritic cells for immunotherapy. Vaccine. 2012 Jan 5;30(2):378-87. doi: 10.1016/j.vaccine.2011.10.081. Epub 2011 Nov 12. PMID 22085546
- [Background] Ten Brinke A, Hilkens CM, Cools N, Geissler EK, Hutchinson JA, Lombardi G, Lord P, Sawitzki B, Trzonkowski P, Van Ham SM, Martinez-Caceres EM. Clinical Use of Tolerogenic Dendritic Cells-Harmonization Approach in European Collaborative Effort. Mediators Inflamm. 2015;2015:471719. doi: 10.1155/2015/471719. Epub 2015 Dec 24. PMID 26819498
- [Background] Bell GM, Anderson AE, Diboll J, Reece R, Eltherington O, Harry RA, Fouweather T, MacDonald C, Chadwick T, McColl E, Dunn J, Dickinson AM, Hilkens CM, Isaacs JD. Autologous tolerogenic dendritic cells for rheumatoid and inflammatory arthritis. Ann Rheum Dis. 2017 Jan;76(1):227-234. doi: 10.1136/annrheumdis-2015-208456. Epub 2016 Apr 26. PMID 27117700
- [Background] Mansilla MJ, Contreras-Cardone R, Navarro-Barriuso J, Cools N, Berneman Z, Ramo-Tello C, Martinez-Caceres EM. Cryopreserved vitamin D3-tolerogenic dendritic cells pulsed with autoantigens as a potential therapy for multiple sclerosis patients. J Neuroinflammation. 2016 May 20;13(1):113. doi: 10.1186/s12974-016-0584-9. PMID 27207486
- [Derived] Willekens B, Presas-Rodriguez S, Mansilla MJ, Derdelinckx J, Lee WP, Nijs G, De Laere M, Wens I, Cras P, Parizel P, Van Hecke W, Ribbens A, Billiet T, Adams G, Couttenye MM, Navarro-Barriuso J, Teniente-Serra A, Quirant-Sanchez B, Lopez-Diaz de Cerio A, Inoges S, Prosper F, Kip A, Verheij H, Gross CC, Wiendl H, Van Ham MS, Ten Brinke A, Barriocanal AM, Massuet-Vilamajo A, Hens N, Berneman Z, Martinez-Caceres E, Cools N, Ramo-Tello C; RESTORE consortium. Tolerogenic dendritic cell-based treatment for multiple sclerosis (MS): a harmonised study protocol for two phase I clinical trials comparing intradermal and intranodal cell administration. BMJ Open. 2019 Sep 9;9(9):e030309. doi: 10.1136/bmjopen-2019-030309. PMID 31501122
- See also: European Cooperation in Science and Technology (COST), Action BM1305 "Action to focus and accelerate cell-based tolerogenic therapies" — http://www.afactt.eu